CLINICAL TRIAL: NCT00557141
Title: AsthmaCare Study Covering Adherence, Drug Use, Will to Take Part in Shared Decisioning in Asthma Outpatients
Brief Title: Observational Study Regarding Adherence, Drug Use, Will to Take Part in Shared Decisioning in Asthma Outpatients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Heidelberg Metasystems GmbH (Industry)
Responsible Party: Dr. Dr. Thomas Froehlich, Heidelberg Metasystems GmbH
Other Study IDs: S-299/2007
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Asthma
Keywords: Single arm observational retrospective and prospective study
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Age > 18 years, Asthma with irregular or regular use of short acting beta-agonists and / or: Asthma treatment with inhaled steroids, Ability to understand the questionnaire

SUMMARY:
In a private practice setting typical for ambulatory medicine in Germany, asthma staging according to the GINA guidelines will be correlated with "real life" treatment and self management of adult outpatients suffering from asthma. Attitudes concerning adherence, awareness, interest in shared decision making and knowledge about the disease are assessed.

DETAILED DESCRIPTION:
The study focuses on outpatients that have two different types of treatment at hand: on-demand reliever treatment and anti-inflammatory treatment. We will assess the correlation of number of devices and medications in regular or intermittent use with doctors recommendations and prescriptions and the parameters adherence, awareness, interest in shared decision making and knowledge about the disease.

The patients will be seen two to three times. The first visit is used to inform the patient about the study, to check with regard to inclusion and exclusion criteria, and finally to sign the informed consent, if the patient agrees to be enrolled in the study. The patient then will get the questionnaire, and she or he is asked to collect all asthma related medications in continuous or intermittent use and to bring them to the private practice staff.

In the second visit, the private practice staff will check the medications the patient has brought. This is a physical check, i.e. it is based on devices and medications on the desk, not on questions.

At least six months later, the private practice staff will check all asthma related prescriptions for the patient concerned, and for the last six months. The patient will be asked to give information if the questionnaire has not been answered completely.

In a previous study with 1.670 paediatric outpatients enrolled we have shown under-diagnosis, under-treatment and a low overall effectiveness of paediatric outdoor patient asthma care. In this previous paediatric study we compared suspected diagnosis and reported treatment. We did not assess parameters indicating low or high adherence, nor did we ask for interest in shared decision making or for awareness and indicators for knowledge about the disease.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Asthma with irregular or regular use of short acting beta-agonists and/or:
* Asthma treatment with inhaled steroids
* Ability to understand the questionnaire

Exclusion Criteria:

* Age < 18 years
* Significant airway disease other than asthma
* Asthma treatment with fixed combination of inhaled steroids with long or short acting beta-agonists
* Ability to understand the questionnaire must be doubted

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care outpatiens of private practices in Germany, Age > 18 years, Asthma with irregular or regular use of short acting beta-agonists and / or: Asthma treatment with inhaled steroids, Ability to understand the questionnaire
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-05 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Number of devices and packages of asthma medication in regular or intermittent individual use per asthma patient at time of enrollment and after an at least six months follow up period | 6 months

SECONDARY OUTCOMES:
patients adherence,patients content with her / his health status and asthma treatment, patients awareness with regard to asthma treatment, interest in shared decision making, self-reported quality of life under asthma treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas . Froehlich, Dr. Dr.med., Principal Investigator — Kaiserstrasse 11 A, D 69115 Heidelberg
Locations (2):
- Germany (2):
  - Weinmann, Steffen, Dr., Bammental, Baden-Wurttemberg
  - Heidelberg Metasystems GmbH, Heidelberg, Baden-Wurttemberg

REFERENCES:
- [Background] Froehlich T, Henningsen P, Miall DS, Paetzold W, Ross A (2001) The Heidelberg Outdor Patient Asthma Study. XXthCongress of the European Academy of Allegology and Clinical Immunology, 9-13 May 2001, Berlin, Germany